CLINICAL TRIAL: NCT03408652
Title: Multicenter Randomized Phase III Study Evaluating the Efficacy and Safety of Systemic Treatments of Bone Metastases From Kidney Cancer in Patients Treated With Targeted Therapies
Brief Title: Efficacy and Safety of Systemic Treatments of Bone Metastases From Kidney Cancer in Patients Treated With Targeted Therapies
Acronym: MOSCAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOSCAR; 2017-004075-31 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Bone Metastases
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): bone targeted treatment (denosumab or zoledronic acid)
  Interventions: Drug: denosumab
- Arm B (No Intervention): no specific treatment

INTERVENTIONS:
Drug: denosumab — Single subcutaneous injection of denosumab 120 mg every 4 weeks One intravenous infusion of zoledronic acid 4 mg every 4 weeks, according to labelled use.
  Other Names: zoledronic acid
  Arms: Arm A

SUMMARY:
Multicenter, randomized, open-label, 2-arm, parallel-group, phase III study whose goal is to assess the efficacy and safety profile of bone-targeted treatments (Arm A: denosumab or zoledronic acid) versus the control arm (Arm B: no specific treatment) in patients with bone metastases under targeted therapy for Metastatic Renal Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically proven mRCC.
* Administration of one of the systemic agents in use for the treatment of mRCC (no more than three prior systemic therapy regimens). Patients with at least 6 months of 1st line treatment and a bone event may be included.
* More than 1 bone metastasis.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
* Adequate renal function (serum creatinine ≤ 200 mmol/L or creatinine clearance ≥ 30 mL/min according to Cockroft formula or MDRD formula for patients older than 65 years).
* Covered by a medical insurance.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Signed informed consent.
* Accepting to use effective contraception during study treatment and within 5 months after final dose of study therapy.

Exclusion Criteria:

* Prior bisphosphonate or denosumab treatment in the year before inclusion.
* Imminent or ongoing nerve or spinal compression as per the investigator's judgement.
* Ongoing first-line therapy, started for less than 6 months (patients with BM at time of metastases diagnosis will initially benefit from the angiogenesis targeted agents used and are not at higher risk).
* Anticancer treatment under investigation.
* Paraneoplastic hypercalcemia (corrected total calcium > 2.7 mmol/L).
* Grade 4 toxicity under previous targeted agents.
* Liver failure (AST and/or ALT ≥ 5.0 x upper limit of normal (ULN) or total bilirubin beyond normal limits).
* Severe hypocalcaemia > 2.8 mmol/l.
* Fructose intolerance.
* Invasive dental procedure (i.e. tooth extraction, dental implants, oral surgery) within the 10 days prior to randomization or required dental procedures at the pre-inclusion dental examination.
* Psychological, familial, sociological, geographical conditions that would limit compliance with study protocol requirements.
* Pregnant or breastfeeding woman. Females of child-bearing potential must have a negative serum pregnancy test within 7 days prior inclusion.
* Life expectancy ≤ 3 months.
* Participation to another clinical trial that might interfere with the evaluation of the main criterion.
* Known hypersensitivity to the active substance or to any of the excipients of bisphosphonate or denosumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Time to first Skeletal Related Event | Up to 54 months after the first inclusion
  Defined as the time from randomization to first SRE. Patients without event will be censored at the time of the last clinical evaluation.

SECONDARY OUTCOMES:
Number of specific event-free survivals | Up to 54 months after the first inclusion
  Specific times from randomization to appearance of the first Skeletal Related Event.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Every 3 months until the 18th month for each patient
  Incidence of adverse events (AEs) assessed using the National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTCAE) v4 grading scale, specific registration of ONJ or other osteonecrosis and rate of skeletal event per patient during study duration
Evolution of pain severity | Every 3 months until the 18th month for each patient
  Proportion of patients with a clinically meaningful change in pain severity evaluated using a numerical rating scale (NRS)
Evolution of pain | Every 3 months until the 18th month for each patient
  Proportion of patients that shifted from not taking a strong opioid at baseline
Patient's condition evaluation | Up to 9 months for each patient (evaluated at baseline, months 3, 6, 9)
  "Functional Assessment of cancer Therapy-General (FACT-G)" questionnaire, made of 27 items measuring the respondents' health state, each of which is answered using a five-point scale from 0 (not at all) to 4 (very much). Questions are phrased so that higher numbers indicate a better health state. Subscale scores are added to obtain total score.
Patient's condition evaluation | Up to 18 months for each patient (evaluated at baseline, months 3, 6, 9 and 18)
  "EuroQoL 5 Dimensions 5 Levels" questionnaire is a scale used in the health state description. Each items is a three-level scale : having no problems, having some or moderate problems, being unable to do/having extreme problems.The respondents are asked to choose one of the statements which best describes their health status of surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Overall survival | Up to 54 months after the first inclusion
  Measured from the date of randomization to the date of death from any cause
Evaluation of the different practices for bone metastases treatments | Up to 18 months for each patient
  Financial evaluation of centers' practices (home or hospitalization)
Cost-utility analysis | Up to 18 months for each patient
  All the hospitalization costs will be collected during the timeframe: outpatient, inpatient, and home care
Cost-effectiveness analyses | Up to 18 months for each patient
  All the hospitalization costs will be collected during the timeframe: outpatient, inpatient, and home care
Budget impact analysis | Up to 18 months for each patient
  Quantification of financial consequences of rolling out this kind of medical supportive care strategy throughout the health system.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie NEGRIER, PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France